CLINICAL TRIAL: NCT07081217
Title: [18F]Radiocaine: Radiation and Radiochemical Safety
Brief Title: Radiocaine Safety Study In Healthy Human Subjects
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Lutroo Imaging LLC (Industry)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LTR-001
Record Dates: First submitted 2025-07-03; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Healthy Subjects
Keywords: Radiocaine; PET imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Healthy subjects (Experimental)
  Interventions: Diagnostic Test: Intravenous Radiocaine

INTERVENTIONS:
Diagnostic Test: Intravenous Radiocaine — Intravenous injection of Radiocaine

SUMMARY:
This is a Phase 1, single-center, open-label study evaluating the safety, biodistribution, and radiation dosimetry of Radiocaine™, an investigational fluorine-18-labeled PET radiotracer designed to bind voltage-gated sodium channels in pain-related peripheral nerves. The study will enroll healthy adult volunteers and aims to inform future clinical development in pain imaging. Radiocaine™ is being developed as a potential imaging biomarker for the localization and quantification of pain.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, open-label study evaluating the safety, biodistribution, and radiation dosimetry of Radiocaine™, an investigational fluorine-18-labeled PET radiotracer designed to bind to voltage-gated sodium channels expressed in peripheral nerves.

The study will enroll six healthy adult volunteers, each of whom will receive a single intravenous dose of Radiocaine™. Serial PET/MR imaging will be performed over several hours post-injection to assess the distribution of the radiotracer in various tissues and organs. Blood and urine samples will be collected at predefined timepoints to support pharmacokinetic and dosimetry modeling. Safety assessments-including vital signs, laboratory tests, and monitoring for adverse events-will be conducted throughout the study.

The primary objectives are to:

* Evaluate the safety and tolerability of a single dose of Radiocaine™ in healthy individuals;
* Characterize the biodistribution of Radiocaine™ in key organs and tissues;
* Estimate radiation exposure (dosimetry) to inform future clinical use.

These data will guide dosing, image acquisition timing, and safety thresholds for upcoming studies in patients with chronic or neuropathic pain. The results will also support the further development of Radiocaine™ as a potential molecular imaging biomarker for the localization and quantification of pain in human subjects.

This study is intended for early-stage characterization of Radiocaine™ in preparation for future clinical studies involving patients.

ELIGIBILITY:
Inclusion Criteria:

* Pain-free
* Unremarkable baseline health without report of chronic or acute pain

Exclusion Criteria:

* Physical pain of almost any severity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Radiation absorbed dose/Effective dose | 1 day
Adverse events | 30 days
  Presence/absence of adverse events

OTHER OUTCOMES:
Biodistribution | 1 day
  Biodistribution of Radiocaine

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided